CLINICAL TRIAL: NCT01781325
Title: Patient Self Monitoring to Transfer Physical Therapy Exercise From Clinic to Home
Brief Title: Patient Self Monitoring of Physical Therapy Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant ended before study could be initiated
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Florence Sheehan, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IBEHR; R21HS021733 (AHRQ)
Record Dates: First submitted 2012-10-12; First posted 2013-02-01 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Patellofemoral Syndrome
Keywords: musculoskeletal, physical therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBEHR (Active Comparator): IBEHR
  Interventions: Device: IBEHR
- Standard therapy (No Intervention): written instructions

INTERVENTIONS:
Device: IBEHR — physical therapy device to educate patients in physical therapy exercise performance
  Arms: IBEHR

SUMMARY:
Our objective is to develop an IBEHR (Image-Based Electronic Health Record) to show patients how to reproduce at home the exercises prescribed by their physical therapist (PT) in clinic. The IBEHR can also record home exercise sessions for review by and feedback from the PT. The HEALTH CARE BENEFITS of the IBEHR for patient self monitoring are: improved transfer of physical therapy exercise from clinic to home, increased adherence to the exercise prescription, and recording home exercise to assist PT decision making.

DETAILED DESCRIPTION:
Our objective is to develop an IBEHR (Image-Based Electronic Health Record) to help patients to transfer and reproduce at home the exercises they were prescribed by their physical therapist (PT) in clinic. More than 17 million (M) patients are diagnosed with conditions that may benefit from PT in the U.S. each year. Adherence to home exercise is the most important factor in functional recovery, and feedback from the exercise prescriber is the most important factor in achieving patient adherence. However in current practice the patient only gets feedback at clinic visits which may be weeks apart.

The proposed IBEHR will give patients visual feedback in real time comparing their performance at each repetition at home with a recording of themselves performing the exercise correctly in the clinic under the PT's supervision. The visual graphics show the patient how to better position his/her body and extremities. Such feedback is likely to improve adherence with the treatment regimen in terms of frequency, duration, and correctness of exercise, and thus facilitates transition of care between clinic and home.

The IBEHR is also a telemedicine tool because the patient can transmit recordings of home exercise to the PT for rapid review and feedback.

A third benefit of the IBEHR is to improve health care decision making by the PT. In current medical practice, it is difficult for a PT to determine why a patient fails to recover as expected. By recording the exercise performed at home, the IBEHR provides monitoring data that informs the PT whether the patient adhered poorly to prescribed exercise frequency or duration, the patient performed the exercise incorrectly, or the PT prescribed the wrong exercise.

Our Specific Aims are to 1) develop the IBEHR software, 2) perform alpha testing of device accuracy and beta testing of user interface ease of use, and 3) perform preliminary evaluation of the efficacy of the IBEHR to improve adherence.

The HEALTH CARE BENEFITS of the IBEHR for patient self monitoring are: improved transfer of physical therapy exercise from clinic to home, increased adherence to the exercise prescription, and recording home exercise to assist PT decision making.

ELIGIBILITY:
Inclusion Criteria:

* anterior knee pain or anterior cruciate ligament (ACL) injury, including non-operative and post-surgical patients

Exclusion Criteria:

* non computer literate
* nonambulatory
* non English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
adherence to physical therapy exercise | 4 to 8 weeks
  frequency (sessions, repetitions) and correctness of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Florence Sheehan, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States